CLINICAL TRIAL: NCT00885898
Title: Out-of-Hospital Non-Invasive Ventilation in Patients With Acute Respiratory Insufficiency
Brief Title: Out-of-Hospital Non-Invasive Ventilation for Patients With Acute Respiratory Failure
Acronym: NIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Göttingen (Other)
Responsible Party: Dr. med. Markus Roessler, M.D., D.E.A.A., EDIC, Dept. of Anesthesiology, Emergency- & Int. Care Med., Univ. Med. Goettingen, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 40/11/04 UGoettingen
Record Dates: First submitted 2009-04-20; First posted 2009-04-22 (Estimated); Last update posted 2009-04-22 (Estimated); Status verified 2009-04

CONDITIONS: Respiratory Insufficiency; Respiratory Failure
Keywords: Respiratory Insufficiency; Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): "Non-invasive ventilation"
  Interventions: Procedure: Non-invasive-ventilation
- 2 (Active Comparator): "Conventional"
  Interventions: Procedure: conventional treatment

INTERVENTIONS:
Procedure: Non-invasive-ventilation — increased oxygen fraction, continuous positive pressure ventilation, if necessary pressure support ventilation or even intermittent positive pressure ventilation
  Arms: 1
Procedure: conventional treatment — oxygen, diuretics, bronchodilators, positive inotropic drugs
  Arms: 2

SUMMARY:
In the past, patients suffering from acute respiratory failure had to be treated with Oxygen and specific medication, or - if this had not been sufficient - had to be anesthesized and had to undergo endotracheal intubation for invasive ventilation. Nowadays, since emergency ventilators are available that can be used for non-invasive ventilation, the purpose of this study is to investigate if non-invasive ventilation is safe, feasible and effective for the treatment of acute respiratory failure and if less patients will need to be intubated out-of-hospital as well as in the further course.

DETAILED DESCRIPTION:
Single center, prospective, randomized, intention-to-treat clinical trial. The study has been performed within a two tier EMS system of a major city. Prehospital emergency physicians are on scene in every patient enrolled to the study.

Patients with acute respiratory failure (SaO2 < 90%, respiratory rate > 20/min) were enrolled to the study using envelopes for randomisation for either "conventional" (O2 + medication) or "NIV." Vital signs have been documented as well as venous blood gases have been taken every 10 minutes after treatment has been started.

Primary endpoints are 28-day mortality, hospital-, ICU- and respirator-days, SAPS, SOFA II and complications. Secondary endpoints are out-of-hospital incidence of invasive ventilation, effect on SpO2, CO2, respiratory rate, heart rate and blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* acute respiratory failure
* at least 18 years old
* cooperative

Exclusion Criteria:

* cardiac arrest
* respiratory arrest
* unconscious
* uncontrollable agitation
* less than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2005-03; Primary Completion 2007-01 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
28-day-mortality, ICU-days, respirator-days, SAPS, SOFA II, complications | 30 days after enrollment

SECONDARY OUTCOMES:
out-of-hospital incidence of invasive ventilation, effect on SpO2, CO2, respiratory rate, heart rate and blood pressure | 30 days after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Markus S Roessler, Dr. med., M.D., D.E.A.A., EDIC, Study Director — Department of Anesthesiology, Emergency- and Intensive Care Medicine, Georg-August-University Goettingen, Germany
Locations (1):
- EMS, Göttingen, Lower Saxony, Germany

REFERENCES:
- [Background] Roessler M. [Non-invasive ventilation in prehospital emergency medicine]. Anasthesiol Intensivmed Notfallmed Schmerzther. 2008 Apr;43(4):264-6. doi: 10.1055/s-2008-1076608. German. PMID 18409119